CLINICAL TRIAL: NCT03267849
Title: Lamina Cribrosa Depth Change With Change in Eye Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Topcon Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00133667
Record Dates: First submitted 2017-08-29; First posted 2017-08-30 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Glaucoma, Open-Angle
Keywords: biomarker
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- persons drinking water (Experimental): all persons in the study will have images of the eye at baseline eye pressure, then the intervention will be to drink 2 bottles of water to increase eye pressure or decrease eye pressure, then will have images taken a second time
  Interventions: Other: wearing swimming goggles or having laser suturelysis

INTERVENTIONS:
Other: wearing swimming goggles or having laser suturelysis — Two images will be compared in each subject at two different eye pressures with the higher pressure having been produced by the interventions

SUMMARY:
This is a study of the compliance of the lamina cribrosa with change in eye pressure.

DETAILED DESCRIPTION:
Glaucoma patients and control subjects will have their internal eye structure (lamina cribrosa) imaged by optical coherence tomography (OCT) standard images at two different eye pressures. In some participants, the eye pressure will be changed by one of two interventions, wearing goggles or having laser suturelysis

ELIGIBILITY:
Inclusion Criteria:

* persons who consent to drink water and be imaged

Exclusion Criteria:

* non-consenting persons
* those who cannot be imaged

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Change in anterior lamina cribrosa depth | Up to 2 months
  OCT position of lamina measured at 2 eye pressures. Data will be calculated as change in parameters of interest per mm Hg change in eye pressure

CONTACTS AND LOCATIONS:
Overall Officials: Harry A Quigley, MD, Principal Investigator — Professor
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
deidentified information (imaging data) will be shared after initial publication
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: after initial publication, indefinitely
Access Criteria: no restrictions

REFERENCES:
- [Derived] Czerpak CA, Kashaf MS, Zimmerman BK, Mirville R, Gasquet NC, Quigley HA, Nguyen TD. The Strain Response to Intraocular Pressure Increase in the Lamina Cribrosa of Control Subjects and Glaucoma Patients. Transl Vis Sci Technol. 2024 Dec 2;13(12):7. doi: 10.1167/tvst.13.12.7. PMID 39630437
- [Derived] Czerpak CA, Quigley HA, Nguyen TD. Long-term Remodeling Response in the Lamina Cribrosa Years after Intraocular Pressure Lowering by Suturelysis after Trabeculectomy. Ophthalmol Glaucoma. 2024 May-Jun;7(3):298-307. doi: 10.1016/j.ogla.2024.01.003. Epub 2024 Jan 24. PMID 38272391
- [Derived] Hannay V, Czerpak CA, Quigley HA, Nguyen TD. A noninvasive clinical method to measure in vivo mechanical strains of the lamina cribrosa by optical coherence tomography. medRxiv [Preprint]. 2023 Aug 16:2023.08.14.23294082. doi: 10.1101/2023.08.14.23294082. PMID 37645852
- [Derived] Czerpak CA, Kashaf MS, Zimmerman BK, Quigley HA, Nguyen TD. The Strain Response to Intraocular Pressure Decrease in the Lamina Cribrosa of Patients with Glaucoma. Ophthalmol Glaucoma. 2023 Jan-Feb;6(1):11-22. doi: 10.1016/j.ogla.2022.07.005. Epub 2022 Jul 19. PMID 35863747